CLINICAL TRIAL: NCT06362200
Title: The Validation and Biological Index Studies on the Improved Social Function of Autism Spectrum Disorder by 40 Hz Transcranial Alternating Current Stimulation
Brief Title: The Validation and Biological Index Studies on the Improved Social Function of ASD by 40 Hz tACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Jian-Jun Ou, Principal investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LYG20230083
Record Dates: First submitted 2024-03-18; First posted 2024-04-12 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 40 Hz tACS group (Experimental): 40 Hz tACS group participants will receive tACS intervention stimulation (40Hz, 2.0mA, 20 minutes per session, three times a day, 21 times in total) for 1 week.
  Interventions: Device: 40 Hz tACS intervention
- control group (Placebo Comparator): the control group will be given the same frequency of pseudo-stimulation (0mA, 20 minutes per session, three times a day, 21 times in total) for 1 week.
  Interventions: Device: 40 Hz tACS intervention

INTERVENTIONS:
Device: 40 Hz tACS intervention — The central electrode is placed in the CP6 and the other four electrodes are placed around the CP6. 40 Hz tACS group participants will receive alternating current stimulation (40Hz, 2.0mA, 20min/time, three times a day, 21 times in total) for 1 week. Subjects in the placebo comparator group will receive sham tACS for 1 week, which mimics the tACS intervention in terms of electrode placement and session frequency. However, the device will deliver a 0mA current, ensuring no actual stimulation occurs.

SUMMARY:
In this proposed study, tACS will be used to intervene in the autism spectrum disorders of children and adolescents, and the efficacy of this intervention method will be evaluated, as well as the internal mechanism of adolescents' autism spectrum disorders will be discussed.

DETAILED DESCRIPTION:
The objective of this clinical study is to investigate the effects and mechanisms of transcranial alternating current stimulation (tACS) on neural modulation in the right temporoparietal junction (rTPJ) of autism spectrum disorders. The primary inquiry it seeks to address is the impact of tACS the treatment of autism spectrum disorders (ASD) through its influence on the rTPJ . Participants will undergo baseline assessments of clinical symptoms and cognitive levels, utilize electroencephalography (EEG) to monitor brain electrical activity during both resting and task states, analyze EEG neurophysiological characteristics, use eye tracking technology to collect data on participants' eye movements during cognitive tasks, employ functional magnetic resonance spectroscopy (fMRS) to detect neurotransmitters such as glutamate + glutamine (Glx), GABA+ macromolecules (GABA+) and taurine in resting state and Theory of Mind task, as well as utilize magnetic resonance imaging (MRI) to detect and analyze functional connectivity and synchronous activation of relevant brain regions during both resting state and task state. Following completion of baseline assessment and examination, participants will be randomly assigned into two groups: a 40 Hz tACS group and a sham stimulation group with 30 patients in each group for a total of 60 patients. Subjects in the tACS group will receive tACS intervention at 2.0mA with a frequency of 40Hz while subjects in the sham group will receive placebo stimulation at a similar location and frequency with no current between periods. Standardized assessment tools along with Theory of Mind tasks will be utilized to evaluate multidimensional changes in clinical symptoms and cognitive levels post-intervention. Additionally, EEG will again be used to monitor brain electrical activity during both resting and task states by analyzing functional E/I values (fE/I) as well as indicators of EEG oscillatory activity such as α- power, γ-power etc., Eye tracker data analysis will also be conducted again for changes in eye fixation during cognitive tasks while fMRS analysis will focus on changes in neurotransmitters. Furthermore, MRI analysis post-intervention aims to examine changes in functional connectivity along with synchronous activation within rTPJ region alongside related brain regions once more. Researchers aim to validate the efficacy & safety profile associated with 40 Hz tACS intervention within rTPJ for treating social impairment observed within ASD population whilst exploring biological indicators & mechanisms underlying effective treatment strategies involving 40 Hz tACS intervention program.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-18 years old.
2. has been clinically diagnosed with autism spectrum disorder by a psychiatrist
3. Meet the diagnostic criteria for ASD recommended by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
4. Consistent with the diagnosis of ASD by used the Autism Diagnostic Interview Tool - Revised Edition (ADI-R) and the Autism Diagnostic Observation Tool (ADOS) assessment.
5. Can cooperate with transcranial alternating current stimulation.

Exclusion Criteria:

b) There is a serious neurological disorder, a clear family history or a potential risk.

c) There are metal implants in the brain, holes or cracks in the skull. e) The presence of a definite or suspected genetic disorder.

1. the presence of common genetic disorders, such as trisomy 21 syndrome
2. The presence of serious physical diseases, such as significant intracranial lesions, thyroid disease, epilepsy, congenital heart disease, severe blood system diseases, systemic lupus erythematosus, audio-visual impairment, etc.
3. meet the diagnosis of other major mental disorders, such as schizophrenia and bipolar disorder.
4. Imaging examination reveals obvious abnormalities in brain structure.
5. Currently taking or have taken benzodiazepine medications or antiepileptic drugs within the past week.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2024-04-07 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Autism assessment assessment index | At baseline, the day after intervention, three weeks after intervention
  Autism was assessed using the Oregon State University Autism Rating Scale, DSM-5 (OARS-5), which includes the signs and symptoms of autism spectrum disorders described in the DSM-5. The scores include :1; Total number of symptoms. Every symptom that occurs (i.e., 1, 2, or 3 points) is recorded in the symptom count. 2. Weighted average severity. The clinician scored each item on a scale of 0, 1, 2 or 3 based on the parent's description of the particular problem. 3. Damage index. In Section C of OARS-5, after discussion with the child/adolescent's caregiver, the clinician will rate the level of support on a scale of 0(no support) to 3(maximum support).

SECONDARY OUTCOMES:
EEG physiological detection index | At baseline, the day after intervention, three weeks after intervention
  detect resting state and task state EEG, analyze and calculate the functional E/I ratio of EEG power spectrum
Magnetic resonance detection index | At baseline, the day after intervention, three weeks after intervention
  Functional magnetic resonance imaging (fMRI) data were used to analyze the functional status and network connectivity between rTPJ and other brain regions. Glx, GABA+, taurine and other neurotransmitters were detected by magnetic resonance spectroscopy to evaluate the changes in the key transmitters of neural E/I balance.
Eye movement index | At baseline, the day after intervention, three weeks after intervention
  Eye tracker was used to record the visual movement trajectories of the subjects when they were performing cognitive tasks, and these movement patterns were analyzed to understand the subjects' attention concentration points and emotional responses in different task situations.
Emotion recognition index | At baseline, the day after intervention, three weeks after intervention
  The "Reading the Mind in the Eyes" test is a psychological assessment to measure subject's ability to understand or infer the mental states of others through the observation of their eyes. It's used to investigate social cognition, empathy, and theory of mind.
Understanding of social interaction index | At baseline, the day after intervention, three weeks after intervention
  The Frith-Happe animations task is used to measure individuals' ability to understand and interpret social interactions. In this task, participants are shown 8 short animated video clips depicting simple social interactions between triangle shapes. Participants will be asked whether the type of interaction of triangles in these animations is random or psychological, and be rated according to their choice of the type of interaction presented by the triangle animation. Each animation gets one point if it chooses the interaction type correctly; otherwise, it gets zero points. The total score is eight.
Understanding of thoughts and intentions index | At baseline, the day after intervention, three weeks after intervention
  Strange Stories Task involves presenting participants with a series of short narrative vignettes that involve interactions between characters that require the reader to infer the characters' thoughts, beliefs, intentions, and emotions. After reading each story, participants are asked questions or prompted to make judgments about the characters' mental states, motivations, and interpretations. Responses are then scored based on the participant's ability to accurately interpret the social cues presented in the narratives. Each question is scored 0, 1, and 2 according to the scoring standard.
Social Communication Changes index | At baseline, the day after intervention, three weeks after intervention
  Assessed by the Social Response Scale (SRS-II). The change in social communication scores from baseline to the end of the study period will be the primary outcome of interest, the critical value is 59.5, and the total score is the sum of all entries, with the lowest score of 0 and the highest score of 3 for each entry.
Stereotyped behavior index | At baseline, the day after intervention, three weeks after intervention
  The Repetitive Stereotyping Behavior Scale-Revised (RBS-R) is a tool used to assess repetitive and stereotyping behaviors in autism spectrum disorders (ASD) and other related disorders. The scale consists of 5 subscales, namely Ⅰ stereotypical behavior scale, Ⅱ self-injury behavior scale, Ⅲ impulsive behavior scale, Ⅳ ritualistic behavior scale, Ⅴ fixed behavior scale, and the score is 0= these behaviors have never happened -- 3= these behaviors have happened. And it's serious; The number of positive items is items other than those with a zero score.
Sensory index | At baseline, the day after intervention, three weeks after intervention
  The Short Sensory Profile (SSP) was used to assess sensory processing abnormalities in children. Each statement has a rating range, which is a 5-point scale from "always" to "never." Raters need to rate the child based on how often they respond to specific sensory inputs. The total score of the SSP is the sum of the scores of all entries. The lowest score generally reflects a higher level of sensory processing difficulty, while the highest score indicates less difficulty.
Abnormal behavior indicator | At baseline, the day after intervention, three weeks after intervention
  Individuals are assessed for behavioral abnormalities using the Aberrant Behavior Checklist-Second Edition (ABC-II), a scoring system designed according to the frequency and severity of behavioral problems. For each entry, raters are asked to rate it according to the following criteria: 0: no problem at all. Score 1: The behavior is problematic, but the degree is not serious. Score 2: The problem is moderately serious. 3 marks: The problem is serious. The total score for ABC-II is the sum of scores for all entries, with the lowest score (i.e., all entries are rated 0) indicating that no behavioral problems were observed, while the highest score (i.e., all entries are rated 3) indicating widespread and serious behavioral problems.
Sleep index | At baseline, the day after intervention, three weeks after intervention
  Childhood Sleep Disorders Scale (SDSC) was used to assess children's sleep problems and habits. Ratings are usually based on frequency and duration, such as "always," "often," "sometimes," "occasionally," or "never happens." Each entry is typically scored on a scale of 0 to 5, with 0 being no problem and the highest being the most serious. The total score of the CSHQ is the sum of the scores of all entries.

OTHER OUTCOMES:
Plasma Metabolite Levels Assessment | At baseline, the first day of intervention
  The levels of metabolites in plasma will be detected and quantified using a comprehensive Metabolomics detection approach. This method involves analyzing small-molecule chemical compounds found in plasma, providing a broad snapshot of the metabolic state of an organism at the given time points.
Safety evaluation SAFTEE indicator | At baseline, the day after intervention, three weeks after intervention
  This scale is the most common safety assessment tool used in clinical trials to assess whether participants experienced side effects or unexpected adverse events during the course of the study. The SAFTEE-GI (General inquiry) version was used in this study, which included detailed inquiry on whether subjects had physical or psychological problems in a specific period of time, occurrence time, duration, occurrence frequency, current status, etc., so as to identify adverse reactions of subjects in the course of clinical trials in a timely manner.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Ou, doctor, Study Chair — Central South University
Locations (1):
- Department of Psychiatry, Xiangya Second Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No